CLINICAL TRIAL: NCT06562660
Title: The Effect of Mask Combined With High Flow Oxygen on Preoxygenation During Induction of General Anesthesia in Obese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HenanPPH-wanghuabing
Record Dates: First submitted 2024-07-28; First posted 2024-08-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Obese
Keywords: High-Flow Nasal Oxygen; Obese Men; Smoking
MeSH Terms: conditions — Obesity; Smoking

STUDY DESIGN:
Intervention Model Description: A total of 60 male obese patients undergoing elective non-thoracic surgery were divided into two groups (n=30) based on smoking status: smokers(S groups), and never smokers(NS groups). Those in the smoking group were current or past smokers, while those in the nonsmoking group had never smoked.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A total of 60 male obese patients undergoing elective non-thoracic surgery were divided into two groups (n=30) based on smoking status: smokers(S groups), and never smokers(NS groups). Those in the smoking group were current or past smokers, while those in the nonsmoking group had never smoked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smoking group (Experimental): In the Smoking group, the HFNC was performed after the patient lost spontaneous breathing until the end-tidal oxygen concentration reached 95 %. record the patient 's safe apnea time.
  Interventions: Device: apnoeic
- never smoking (No Intervention): no intervention

INTERVENTIONS:
Device: apnoeic — In group S, High-Flow Nasal Oxygen was performed after the patient lost spontaneous breathing until the end-expiratory oxygen concentration reached 95 %.
  Arms: Smoking group

SUMMARY:
There is a risk of airway-related incidents during anaesthesia associated with obesity. High-flow nasal oxygen is advocated for perioperative preoxygenation in obese patients to reduce airway adverse reactions. However, there have been no reports on whether smoking behaviors have an impact on obese men's Apnoeic oxygenation with high-flow nasal.This study compared the effects of smoking on the duration of safe apnoea times in obese males.

DETAILED DESCRIPTION:
All patients were were divided into two groups based on smoking status: smokers(S groups), and never smokers(NS groups). Those in the smoking group were current smokers, while those in the nonsmoking group had never smoked. Both groups of patients were induced with intravenous anesthesia and received 5 minutes of high flow nasal oxygen (60 L min) prior to induction.After induction of anaesthesia, the patients were apnoeic until peripheral oxygen saturation decreased to 95 %.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ranged in age from 18 to 80 with BMI≥30 kg/m2.
2. Participants are male obese patients undergoing elective non-thoracic surgery

Exclusion Criteria :

1. patients were kept awake during the intubation due to cervical spine pathology.
2. Patients with unstable hemodynamics.
3. Patients with airway inflammatory diseases, including asthma, chronic obstructive pulmonary disease (COPD), lung cancer, pulmonary fibrosis and cystic fibrosis.
4. Patients with upper respiratory infection and nasal blockage.
5. Patients with Hypersensitivity to the drug.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
the safe apnoea times | 5-minute
  Investigators will record the time of oxygen saturation drop to 95 % during intubation.

SECONDARY OUTCOMES:
the Pao2 levels | 5-minute
  the Pao2 levels after 5-minute pre oxygenation with high flow nasal oxygen in two groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: jiaqiang zhang, Study Director — Chief physician
Locations (1):
- Wanghuabing, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No